CLINICAL TRIAL: NCT03991767
Title: Implementation and Evaluation of an Electronic Alert to Encourage Targeted Screening for HIV Infection at Foch Hospital According to Socio-demographic Criteria: Pilot Study
Brief Title: Implementation and Evaluation of an Electronic Alert to Encourage Targeted Screening for HIV Infection at Foch Hospital According to Socio-demographic Criteria
Acronym: POP-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2016/51
Record Dates: First submitted 2019-06-11; First posted 2019-06-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: HIV Testing
Keywords: medical practices; HIV; Electronic Alert
MeSH Terms: interventions — AIDS Serodiagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- period 1 (Experimental): Period 1: Retrospective period:
  Collection of data from the 12 months preceding the start of the research of hospitalized patients:
  * number of hospitalizations,
  * number of HIV serologies performed,
  * number of patients with socio-demographic criteria justifying HIV screening.
  Start of research: Implementation of the "POP-UP" electronic alert
  Period 2: Prospective period: 18 months POP-UP opens for patient who meet the eligibility criteria.
  Six possibility to answer:
  1. Patient accept to participate: patient is include and receive HIV serology during their hospitalization.
  2. Not time to answer to the alert
  3. Patient already has a serology less than 3 months old
  4. Patient followed for a known HIV infection.
  5. Patient who refused the test
  6. Clinical condition of the patient not allowing his no opposition Only choice 1 include patient The response close the electronic alert, but it re-opens when the medical file is re-consulted (2/ and 6/) or new hospitalization.
  Interventions: Other: "POP-UP" electronic alert; Diagnostic Test: Serology HIV

INTERVENTIONS:
Other: "POP-UP" electronic alert — Implementation of the "POP-UP" electronic alert for all patients with eligibility criteria
Diagnostic Test: Serology HIV — Realization of HIV serology for included patients.

SUMMARY:
In 2013 in France, 29,000 people are reported to be unaware of their HIV status. HIV testing is a priority in France where one third of all diagnoses remain late despite 5 million annual tests. It is recommended to offer at least one HIV test to the general population, over the life course, when seeking care and more frequently to populations at risk. Several international and national articles have shown that emergency screening is feasible and well accepted. But also that during systematic screening few infections were discovered, and the majority of newly diagnosed people belonged to the most exposed groups.

Our hypothesis is that an electronic alert would identify people who are unaware of their HIV status. This alert would be based on two data: social data (French health coverage) and the country of birth. This alert is only relevant in high-prevalence regions, as is the case in the Ile de France region.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized at Foch Hospital over 18 years of age.
* Patient with AME or CMU and/or CMUc, or patient born in one of the following countries/regions: Sub-Saharan Africa, Haiti, South America, Asia, Eastern Europe, Guadeloupe, Martinique and Guyana

Exclusion Criteria:

* Patient whose vital prognosis at the time of admission does not allow him/her to indicate his/her non-opposition to an HIV test.
* Patient being followed for a known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of HIV testing practices : screening proposal rate, patient acceptance rate and serological achievement rate | 18 months
  Evaluation of the practice of hospital doctors at Foch Hospital following the implementation of "POP-UP" electronic alert to encourage targeted screening for HIV infection according to specific socio-demographic criteria :
  * Screening proposal rate (= number of proposition compared to number of eligible patients).
  * Patient acceptance rate (= number of eligible patients acceptances compared to number of screening proposals).
  * Serological achievement rate (= number of serologies compared to number of eligible patients).

SECONDARY OUTCOMES:
Study of the obstacles | 18 months
  Study of the obstacles encountered by clinicians in proposing screening tests induced by electronic alerting by questionnaire of satisfaction.
Prospective data vs retrospective data : number of screening serologies performed | 18 months
  Comparison of the number of screening serologies performed in eligible inpatients by the POP-UP" electronic alert versus the retrospective data of the 12 months preceding the implementation of the alert .
Newly HIV+ | 18 months
  Number of hospitalized patients newly diagnosed HIV
Positivity rate | 18 months
  Number of newly diagnosed HIV vs the number of serologies performed

CONTACTS AND LOCATIONS:
Overall Officials: David Zucman, MD, Study Director — FOCH Hospital
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No